CLINICAL TRIAL: NCT03781986
Title: A Multicenter Phase I/II Trial of a Novel MDM2 Inhibitor (APG-115) in p53 Wild-type Salivary Gland Carcinoma
Brief Title: APG-115 in Salivary Gland Cancer Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.127; APG-115SG101 (Other: Ascentage Pharma); HUM00155822 (Other: University of Michigan IRB)
Record Dates: First submitted 2018-12-06; First posted 2018-12-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Malignant Salivary Gland Cancer; Salivary Gland Cancer
Keywords: p53 wild-type; Adenoid cystic carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic | interventions — Carboplatin

STUDY DESIGN:
Intervention Model Description: Part 1 -- Parallel assignment [terminated early]:
  * Arm A: APG-115 Monotherapy
  * Arm B: APG-115 + Carboplatin
  Part 2 -- Single arm (Arm A only): APG-115 Monotherapy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APG-115 monotherapy (Experimental): APG-115 will be administered in an open label fashion until progression, intolerance, or patient preference.
  Interventions: Drug: APG-115
- APG-115 + Carboplatin [terminated] (Experimental): APG-115 and Carboplatin will be administered in an open label fashion until progression, intolerance, or patient preference. [Phase 1 was terminated early and this arm was discontinued. An MTD was not established during Phase 1.]
  Interventions: Drug: APG-115; Drug: Carboplatin

INTERVENTIONS:
Drug: APG-115 — APG-115 at 150mg (or lower, if dose is reduced) is taken orally every other day through day 13 of each cycle. Cycle length 21 days.
Drug: Carboplatin — Carboplatin is given IV at AUC=4.5 on day 1 of each cycle. Cycle length 21 days.
  Arms: APG-115 + Carboplatin [terminated]

SUMMARY:
This is a phase I/II trial to evaluate the efficacy of APG-115 +/- Carboplatin for the treatment p53 wild-type malignant salivary gland cancer.

Part 1 consisted of 2 arms, arm A (APG-115 monotherapy) and arm B (APG-115 + Carboplatin) and was terminated early.

Part 2 is a single arm study (APG-115 monotherapy).

DETAILED DESCRIPTION:
The current single arm study design was originally part of a study with a parallel arm given combination APG-115 + Carboplatin. In the initial phase of that previous iteration, the combination arm was closed early for issues related to tolerability of the combination therapy. This study will continue as a single arm, monotherapy alone, Phase I/II study as approved by the UM Institutional Review Board as of June 2021.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented malignant salivary gland cancers (including secretory glands of the aerodigestive tract) with or without metastases, not amenable to curative treatment; or there is documentation of patient refusal of curative treatment.
* Previous mutational testing with no evidence of a p53 mutation
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Presence of measurable disease by CT scan per RECIST v1.1 with ≥ 20% increase in tumor burden in the preceding 12 months
* Life expectancy of ≥12 weeks
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Patients must be able to take oral medication without breaking/opening, crushing, dissolving, or chewing capsules
* Adequate organ and marrow function obtained ≤ 2 weeks prior to enrollment

Exclusion Criteria:

* Prior treatment with MDM2 inhibitors
* Patients are not eligible if they have received any systemic anti-cancer therapy (including chemotherapy and/or hormone therapy) for salivary gland cancer within 4 weeks of the start of study therapy
* Patients are not eligible if they have received any of the following within 4 weeks of the start of study therapy: live vaccines, antiretroviral drugs
* Progressive disease within 6 months of the last dose of platinum-based chemotherapy
* Patients with active brain metastases are excluded because of unknown penetration into the central nervous system (CNS). A confirmatory scan for asymptomatic patients is not required. Patients with a history of treated CNS metastases are eligible provided they meet all of the following criteria: disease outside the CNS is present, no clinical evidence of progression since completion of CNS-directed therapy, minimum 4 weeks between completion of radiotherapy and enrollment, and recovery from significant (Grade ≥ 3) acute toxicity.
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment
* Patients (male and female) having procreative potential who are not willing or not able to use 2 adequate methods of contraception or practicing abstinence during the study and for 90 days following their last dose of treatment
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Toxicity Endpoint: dose-limiting toxicity (DLT) | 42 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 6 weeks (2 cycles) of study treatment. These will be assessed via CTCAE version 5.0
Maximally tolerated dose (MTD) | 42 days
  MTD will be determined based on DLTs observed during the first 6 weeks (2 cycles) of study treatment.
Overall response rate | up to 12 months
  Overall response rate will be defined as the proportion of patients achieving either complete response (CR) or partial response (PR). Response will be assessed via RECIST v1.1.

SECONDARY OUTCOMES:
Overall response rate by tumor histology | Until death or end of study; up to approximately 5 years
  Overall response rate will be defined as the proportion of patients achieving either complete response (CR) or partial response (PR), assessed via RECIST v1.1 and reported separately for those with histologically confirmed adenoid cystic carcinoma (ACC) versus other malignant salivary gland tumors (non-ACC)
Duration of response | Until death or end of study; up to approximately 5 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.
Progression-free survival | Until death or end of study; up to approximately 5 years
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever is earlier.
Overall survival | Until death or end of study; up to approximately 5 years
  Overall survival (OS) is defined as the duration of time from start of treatment to time of death or end of study.
Disease control rate | Until death or end of study; up to approximately 5 years
  Defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD). Response will be assessed via RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Swiecicki, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No